CLINICAL TRIAL: NCT03839121
Title: BIO|REDUCE: Cardiac REsynchronization Therapy With Two Ventricular Leads and Right Atrial Floating Diagnostic Dipole Installed in the Right ventricUlar Lead in Patients With CRT-D indiCation and no Sinus nodE Dysfunction
Brief Title: Safety and Performance Aspects of CRT-DX System in Patients With Sinus Rhythm
Acronym: BIO|REDUCE
Status: Completed | Type: Observational
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Other Study IDs: CR024
Record Dates: First submitted 2019-01-11; First posted 2019-02-15 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2022-03

CONDITIONS: Heart Failure; Cardiac Resynchronization Therapy
Keywords: Heart Diseases; CRT-D
MeSH Terms: conditions — Heart Failure; Heart Diseases | interventions — Cardiac Resynchronization Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- single arm: CRT-DX
  Interventions: Device: Cardiac Resynchronization Therapy (CRT)

INTERVENTIONS:
Device: Cardiac Resynchronization Therapy (CRT) — Observation and documentation of CRT patients

SUMMARY:
The conventional CRT-D system consists of 3 leads in patients with Heart Failure (HF). A part of HF patients have non-impaired sinus node function and will not be stimulated in the right atrium. The implantation of the right atrial lead, which is not mandatory in these patients, harbors potential complication risks and prolongs implantation procedure. The new CRT-DX system uses 2 leads only: a right ventricular lead extended with floating RA sending dipole and a left ventricular lead. The aim of the BIO|REDUCE study is to assess the residual safety and performance aspects of the CRT-DX system within 12 months follow-up in HF patients with an indication for a CRT-D, sinus rhythm, and no need for an atrial lead implantation.

ELIGIBILITY:
Inclusion Criteria:

* Patient is able to understand the nature of study and has provided written informed consent.
* Patient is willing and able to perform all follow up visits at the study site.
* Patient is willing and able to use the CardioMessenger® and accepts the BIOTRONIK Home Monitoring® concept.
* CRT-D is indicated according to the current ESC guidelines.
* De novo implantation with no pre-existing defibrillator or pacemaker system
* Patient is in sinus rhythm without history of persistent or permanent atrial fibrillation.
* Patient has no atrioventricular (AV) block II or III.
* Patient has no evidence of impaired sinus node function.
* Patient has no need for atrial stimulation, has a resting heart rate (HR) > 40 b.p.m and achieves a peak HR ≥100 b.p.m even under intended dosage of HR lowering medication verified by an appropriate method as clinical routine examination within 3 months prior to enrollment
* NYHA class II or III
* Patient receives guideline-based optimized medical therapy for HF including heart-rate lowering medication at the time of enrollment

Exclusion Criteria:

* Patient is pregnant or breast feeding.
* Patient is less than 18 years old.
* Patient is participating in an interventional clinical investigation.
* Life-expectancy is less than 1 year.
* Patient has tachycardia-bradycardia syndrome
* Any standard contraindication for CRT-D
* Frequent premature ventricular contractions (PVC rate > 5 %/h) examined within 3 months prior to enrollment by appropriate routine method (e.g. 24 h holter electrocardiogram)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Cardiac Resynchronization Therapy Defibrillator (CRT-D) indication according to the current guidelines, who are in sinus rhythm without history of persistent or permanent atrial fibrillation (AF) and do not require right atrial (RA) lead implantation at study enrolment.
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2023-06-08 (Actual); Study Completion 2023-06-08 (Actual)

PRIMARY OUTCOMES:
Number of implantation of a right atrial lead after conclusion of the initial study device implantation | through study completion, on average 12 months

SECONDARY OUTCOMES:
Number of post-operative system revisions requiring an invasive re-intervention | through study completion, on average 12 months
Number of lead complications requiring an invasive re-intervention | through study completion, on average 12 months
Number of device or pocket infections requiring an invasive re-intervention | through study completion, on average 12 months

OTHER OUTCOMES:
Documentation of patient characteristics and medication | through study completion, on average 12 months
Assessment of patients benefit from CRT | Baseline, 3, 6 and 12 months
  Documentation of NYHA class
Echocardiographic changes - LVEF | Baseline, 6 and 12 months (optional at other visits)
  Echocardiography (measurements of Left ventricular ejection fraction [%] )
Echocardiographic changes - LVESV/LVEDV | Baseline, 6 and 12 months (optional at other visits)
  Echocardiography (optional measurements Left ventricular end-systolic/diatolic volume [ml])
Echocardiographic changes - LVESD/LVEDD | Baseline, 6 and 12 months (optional at other visits)
  Echocardiography (optional measurements Left ventricular end-systolic/diastolic diameter [mm])
Echocardiographic changes - LAV | Baseline, 6 and 12 months (optional at other visits)
  Echocardiography (optional measurements Left atrial volume [ml])
Documentation of atrial sensing amplitude | through study completion, on average 12 months
Documentation of programming of a non-AV-sequential pacing mode (e.g. VVI) except if justified by atrial fibrillation | through study completion, on average 12 months
Documentation of implantation data | through study completion, on average 12 months
  e.g. implantation time, x-ray exposure time, lead position
Number of serious adverse events | through study completion, on average 12 months
  Documentation of serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Christof Kolb, Prof., Principal Investigator — DHM, München
Locations (21):
- Kepler University Clinic, Linz, Austria
- Czechia (2):
  - Fakultni Nemocnice Hradec Králové, Králová
  - Fakultni Nemocnice Olomouc, Olomouc
- Germany (17):
  - RHÖN-KLINIKUM Campus Bad Neustadt, Bad Neustadt an der Saale
  - Vivantes Humboldt-Klinikum, Berlin
  - Herzzentrum Dresden Univesity Clinic at Technical University Dresden, Dresden
  - Städtisches Klinikum Dresden, Friedrichstadt, Dresden
  - Heinrich-Heine University Düsseldorf, Düsseldorf
  - University Clinic Erlangen, Erlangen
  - Elisabeth-Krankenhaus Essen, Essen
  - Westpfalz-Klinikum, Kaiserslautern
  - University Clinic SH Campus Kiel, Kiel
  - Clinic St. Georg, Leipzig
  - DHM, Munich
  - Rheinlandklinikum Neuss GmbH -Lukaskrankenhaus Neuss, Neuss
  - Marien Hospital Papenburg Aschendorf, Papenburg
  - Cardio Consil GmbH, Rostock
  - Krankenhaus Rothenburg ob der Tauber, Rothenburg upon Tauber
  - Charitè University Clinic, Campus Benjamin Franklin, Steglitz
  - University Clinic Würzburg, Würzburg
- Semmelweis Medical University, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: Undecided